CLINICAL TRIAL: NCT05949580
Title: Study to Evaluate the Usability of Introducing Integrated Digital Solutions Into Clinical Practice and the Value of Their Use in the Medical Care of Patients With Multiple Sclerosis (MS)
Brief Title: Study to Evaluate the Usability and Value of Integrated Digital Solutions in Medical Care of Participants With Multiple Sclerosis
Acronym: ILLUMINATE
Status: Recruiting | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: icometrix (Industry)
Responsible Party: Sponsor
Other Study IDs: MN44358
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: icobrain; icompanion; Multiple Sclerosis; Medical device; Patient app; Digital; Care management; Magnetic resonance imaging (MRI); Deep learning; Artificial Intelligence (AI); Patient Reported Outcomes (PRO)
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- People with RRMS: Participants with relapsing-remitting multiple sclerosis (RRMS) will have to complete various questionnaire from which data will be collected for patient-reported outcomes (PROs) using the icompanion patient app and the HCPs will complete various questionnaires using the icompanion HCP portal.
  Interventions: Device: MS Care Platform (icobrain ms and icompanion ms)

INTERVENTIONS:
Device: MS Care Platform (icobrain ms and icompanion ms) — The MS care management platform consists of the following components:
  1. icobrain ms which is a a cloud-based solution to quantify brain volume and brain abnormalities and changes thereof on MRI scans;
  2. icompanion ms which consists of free participant mobile application (app) and a web portal for HCPs.
  The information collected in the icompanion ms patient app and icobrain ms is then brought together in the icompanion ms HCP web portal which allows a comprehensive overview of disease data for every single participant.

SUMMARY:
The main purpose of this study is to assess the usability and value of the multiple sclerosis (MS) care management platform in terms of improved monitoring of people with MS (pwMS) in clinical practice.

This is a two-year prospective data collection study with additional data collection at baseline evaluating medical practice over a period of at least one year before the introduction of the MS care management platform.

DETAILED DESCRIPTION:
The MS care management platform consists of:

A) icobrain ms, a cloud-based artificial intelligence (AI) solution to quantify brain volume and brain abnormalities and changes thereof on magnetic resonance imaging (MRI) scans and thereby providing insights into subclinical changes during disease progression in MS.

B) icompanion ms, which consists of i) A free participant mobile application (app) and website to keep track of participant reported health and medications and prepare participants for the next consultation.

ii) A web portal for healthcare professionals (HCPs), which is accessible via web browser. The MS care team will be able to access the participants' data entered via the participant app (active linking of systems by the participant required), as well as their participants' MRI images and icobrain ms volumetric brain reports automatically imported by the hospital picture archiving and communications system (PACS).

ELIGIBILITY:
Inclusion Criteria:

* Able to comply with the study protocol, including having a smartphone and being able and willing to access the icompanion ms patient app on a regular basis. To use all functionalities of the icompanion ms patient app, the user's smartphone must comply with the minimum system requirements (Android version 5.0 or above, iOS version 11 or above)
* Have a valid email address (for registration of icompanion ms)
* Have a definite diagnosis of RRMS
* Time since MS diagnosis ≥1 year
* Medical history recorded for at least 1 year before enrollment
* Expanded Disability Status Scale (EDSS) <5.5

Exclusion Criteria:

* Any contra-indications to using icompanion ms patient app or website, as per the investigator's discretion
* Inability to complete an MRI
* Currently involved in an interventional trial
* Diagnosis of progressive MS (primary progressive multiple sclerosis [PPMS] or secondary progressive multiple sclerosis [SPMS])

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with MS are enrolled in this study. Participants with RRMS were chosen because most available disease modifying therapies (DMTs) are approved for this subgroup, and hence guiding care in this population is most relevant.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
HCPs: Median of the System Usability Scale (SUS) Score Reported by Radiologists and Neurologists at Month 6 | Month 6
  SUS is a validated scale that assesses subjective usability of a system, or, in this case, the MS care management platform. The SUS consists of a 10-item questionnaire with five response options ranging from Strongly agree (5) to Strongly disagree (1). The items scores are converted into a score from 0 (negative) to 100 (positive). A score of ≥50 indicates that the MS care management platform is acceptable, and a score above 68 is considered above average. The final SUS score is not a percentile or a percentage and the SUS acceptability guidelines on how to interpret the score are: <51=awful; 51-68=poor; 68=okay; 68-80.3=good; > 80.3=excellent; 100=best imaginable score.
HCPs: Median of the SUS Score Reported by Radiologists and Neurologists at Month 12 | Month 12
  SUS is a validated scale that assesses subjective usability of a system, or, in this case, the MS care management platform. The SUS consists of a 10-item questionnaire with five response options ranging from Strongly agree (5) to Strongly disagree (1). The items scores are converted into a score from 0 (negative) to 100 (positive). A score of ≥50 indicates that the MS care management platform is acceptable, and a score above 68 is considered above average. The final SUS score is not a percentile or a percentage and the SUS acceptability guidelines on how to interpret the score are: <51=awful; 51-68=poor; 68=okay; 68-80.3=good; > 80.3=excellent; 100=best imaginable score.
HCPs: Median of the SUS Score Reported by Radiologists and Neurologists at Month 24 | Month 24
  SUS is a validated scale that assesses subjective usability of a system, or, in this case, the MS care management platform. The SUS consists of a 10-item questionnaire with five response options ranging from Strongly agree (5) to Strongly disagree (1). The items scores are converted into a score from 0 (negative) to 100 (positive). A score of ≥50 indicates that the MS care management platform is acceptable, and a score above 68 is considered above average. The final SUS score is not a percentile or a percentage and the SUS acceptability guidelines on how to interpret the score are: <51=awful; 51-68=poor; 68=okay; 68-80.3=good; > 80.3=excellent; 100=best imaginable score.
Participants: Median Score of the mHealth App Usability Questionnaire (MAUQ) [MAUQ_E (Ease of Use) MAUQ_I (Interface and Satisfaction)] at Baseline | Baseline
  MAUQ_E and MAUQ_I are subscales of a validated self-report survey (MAUQ) in which participants report how easy the app (icompanion MS patient app) was to use and rate their satisfaction with the user interface of the app. MAUQ_E consists of a 5-item questionnaire with seven response options ranging from Strongly agree to Strongly disagree. Ease of use scores range from 5 to 35 with higher scores indicating greater ease of use. MAUQ_I consists of a 7-item questionnaire with seven response options; from Strongly agree to Strongly disagree. Interface and satisfaction scores range from 7 to 49 with higher scores indicating greater satisfaction.
Participants: Median Score of the MAUQ (MAUQ_E and MAUQ_I) at Month 12 | Month 12
  MAUQ_E and MAUQ_I are subscales of a validated self-report survey (MAUQ) in which participants report how easy the app (icompanion MS patient app) was to use and rate their satisfaction with the user interface of the app. MAUQ_E consists of a 5-item questionnaire with seven response options ranging from Strongly agree to Strongly disagree. Ease of use scores range from 5 to 35 with higher scores indicating greater ease of use. MAUQ_I consists of a 7-item questionnaire with seven response options; from Strongly agree to Strongly disagree. Interface and satisfaction scores range from 7 to 49 with higher scores indicating greater satisfaction.
Participants: Median Score of the MAUQ (MAUQ_E and MAUQ_I) at Month 24 | Month 24
  MAUQ_E and MAUQ_I are subscales of a validated self-report survey (MAUQ) in which participants report how easy the app (icompanion MS patient app) was to use and rate their satisfaction with the user interface of the app. MAUQ_E consists of a 5-item questionnaire with seven response options ranging from Strongly agree to Strongly disagree. Ease of use scores range from 5 to 35 with higher scores indicating greater ease of use. MAUQ_I consists of a 7-item questionnaire with seven response options; from Strongly agree to Strongly disagree. Interface and satisfaction scores range from 7 to 49 with higher scores indicating greater satisfaction.
Change From Baseline in Perception of Disease Worsening by HCPs, Assessed by Semi-structured Interviews (SSIs) at Month 6 | Baseline to Month 6
  To assess the change in perception of disease worsening by the HCPs, two versions of the SSIs are available, one version is for radiology and the other for neurology. The HCPs are required to answer a set of 3 questions with 6 response options ranging from strongly disagree to strongly agree and also select the reasons for agreeing/disagreeing from the options listed. If HCPs agree, they can select between aspects of the disease activity/progression for which the system provides an increased ability to detect changes. The questionnaire also includes an item with a yes/no response. A scale ranging from 1 to 6 will be attributed to these responses (with 1 being strongly disagree and 6 being strongly agree). The higher the score, the higher the impact of the tools in the perception of disease worsening.
Change From Baseline in Perception of Disease Worsening by HCPs, Assessed by SSIs at Month 12 | Baseline to Month 12
  To assess the change in perception of disease worsening by the HCPs, two versions of the SSIs are available, one version is for radiology and the other for neurology. The HCPs are required to answer a set of 3 questions with 6 response options ranging from strongly disagree to strongly agree and also select the reasons for agreeing/disagreeing from the options listed. If HCPs agree, they can select between aspects of the disease activity/progression for which the system provides an increased ability to detect changes. The questionnaire also includes an item with a yes/no response. A scale ranging from 1 to 6 will be attributed to these responses (with 1 being strongly disagree and 6 being strongly agree). The higher the score, the higher the impact of the tools in the perception of disease worsening.
Change From Baseline in Perception of Disease Worsening by HCPs, Assessed by SSIs at Month 24 | Baseline to Month 24
  To assess the change in perception of disease worsening by the HCPs, two versions of the SSIs are available, one version is for radiology and the other for neurology. The HCPs are required to answer a set of 3 questions with 6 response options ranging from strongly disagree to strongly agree and also select the reasons for agreeing/disagreeing from the options listed. If HCPs agree, they can select between aspects of the disease activity/progression for which the system provides an increased ability to detect changes. The questionnaire also includes an item with a yes/no response. A scale ranging from 1 to 6 will be attributed to these responses (with 1 being strongly disagree and 6 being strongly agree). The higher the score, the higher the impact of the tools in the perception of disease worsening.

SECONDARY OUTCOMES:
Change From Baseline in Time Needed for MRI Review, Assessed by SSIs of Radiologists | Baseline, 6, 12 and 24 months
  To assess the change in time required for MRI review, the radiologists are required to answer a set of 2 questions; one question with a yes/no response (whether icobrain ms save time when reading an MRI) and another question where in the HCPs will express the time saved in minutes (absolute) and in percentage (relative) while reading an MRI while using icobrain ms.
Change From Baseline in Time Needed for Visit Preparation, Assessed by SSIs of Neurologists | Baseline, 6, 12 and 24 months
  To assess the change in time required for visit preparation, the neurologist is required to answer a set of 3 questions with 6 response options ranging from strongly disagree to strongly agree and if the response selected is "agree" a free text field is available to explain the reason for agreeing.
Change From Baseline in Health Literacy Assessed by the Health Literacy Questionnaire (HLQ) | Baseline, 12 and 24 months
  The HLQ explores dimensions of health literacy such as social support relationship with caregivers, health information evaluation or ability to engage with caregivers. Participants will be asked to rate "How strongly do you disagree or agree with the following statements?". The options provided are: strongly disagree, disagree, agree and strongly agree, which are scored from 1 to 4, respectively. In 2nd part of the HLQ, participants will be asked "How easy or difficult are the following tasks for you to do now?" The options for these scales are: cannot do, usually difficult, sometimes difficult, usually easy and always easy, which were scored from 1 to 5, respectively. For both the parts higher the score higher is the health literacy of a participant.
Change From Baseline in Participant Autonomy Assessed by the Patient Activation Measure® 13 (PAM13) | Baseline, 12 and 24 months
  PAM 13 is a measure used to assess the participant knowledge, skill, and confidence for self-management of health, consisting of 13 questions. Each of the 13 items can be answered with one of four possible response options, which are "disagree strongly" (1), "disagree" (2), "agree" (3), "agree strongly" (4). Scores will be summed to calculate the overall raw score, then transformed to a scale with a theoretical range 0 to 100, based on calibration tables, with higher PAM scores indicating higher participant activation.
Change From Baseline in Medication Adherence, Assessed by the Morisky Medication Adherence Scale (MMAS) | Baseline, 12 and 24 months
  The MMAS 8-item questionnaire is a recognized indicator of medication adherence, consisting of 8 questions with a sum score ranging between 0 and 8 points. The higher score indicates higher adherence to the prescribed therapy recommendation. It has been agreed that the score of 8 could be categorized as having high adherence, score between 6 and 7 as medium adherence and scores of 5 and less as low adherence. A positive change score will reflect an improvement in the adherence.
Time in Days Needed for the Successful Installation and Integration of all Components in the MS Care Management Platform | Baseline
Number of HCPs at Each Study Center Registered on the MS Care Management Platform | Up to 24 months
Factors Influencing HCPs Adoption to MS Care Management Platform Measured by SSIs | Baseline, 6, 12 and 24 months
  Factors influencing HCPs adoption to the MS care platform will be measured using the SSIs. The questionnaire includes three items with a yes/no response along with a free text field to provide an elaboration based on the responses selected.
Number of MRI Scans per Study Center Analyzed With icobrain ms | Baseline, 6, 12, 18 and 24 months
Level of Engagement on Platform Assessed Monthly by the Number of Logins and Time Spent on Individual Portal Pages in the HCP Portal | Up to 24 months
Factors Influencing HCPs Adherence Measured by SSIs | Baseline, 6, 12 and 24 months
  Factors influencing HCPs adherence to the MS care platform will be measured using the SSIs. The questionnaire includes three item with a yes/no response along with a free text field to provide an elaboration if 'yes' is selected.
Number of Participants at Each Study Center That Register for the icompanion ms Patient app | Up to 24 months
Reasons for not Registering for icompanion ms Patient app as Described by the HCP Through the icompanion ms HCP Portal | Up to 24 months
Average Number of Activities in the icompanion ms Patient app per Patient per Month | Up to 24 months
Number of Participants Using the icompanion ms Patient app With at Least 2 Activities Within 2 Months, Assessed per Month | Baseline up to 2 months of enrollement (Up to approximately 12 months)
Number of Participants That Stop Using the icompanion ms Patient app (no Activity for More Than 4 Months), Assessed per Month | Up to 24 months
Reasons for not Using the icompanion ms Patient app Regularly as Described by HCP Through the icompanion ms HCP Portal | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — icometrix
Locations (5):
- United States (3):
  - Minneapolis Clinic of Neurology, Golden Valley, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Jersey Shore University Medical Centre, Neptune City, New Jersey
- Germany (2):
  - Universitaetsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - Praxis Dr. med. Max Deist und Michael Ernst ?Sinsheim, Sinsheim

IPD SHARING:
Plan to Share IPD: No
At this stage of our research, we do not intend to share externally individual patient-level data generated by this study. Nonetheless, it remains our objective to ensure the dissemination of our collective insights and findings from the study to the scientific and medical community. All external publications will be appropriately agreed upon by the study collaborators and coordinated as per our publication plan.